CLINICAL TRIAL: NCT05125172
Title: Focus of Attention Effect on Sit to Stand Symmetry in Individuals Post Stroke: A Randomized Cross-over Trial.
Brief Title: Focus of Attention Effect on Sit to Stand Symmetry in Individuals Post Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Western Carolina University (Other)
Responsible Party: Principal Investigator, Ashley Hyatt, Assistant Professor, Western Carolina University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1799540-1
Record Dates: First submitted 2021-10-06; First posted 2021-11-18 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Stroke
Keywords: Motor learning; Focus of attention; Sit to stand
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Randomized cross-over study. Participants will be randomized into the internal or external focus of attention group and one week later they will complete the opposite protocol.
Who Masked: Participant
Masking Description: Participants will not be aware of their group allocation compared to the other group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internal focus of attention group (Active Comparator): Participants will be given instructions that make them think about their body's movements.
  Participants will complete the external focus group second in the cross over.
  Interventions: Other: Focus of Attention
- External focus of attention group (Experimental): Participants will be given instructions that make them think about an outside target or outcome.
  Participants will complete the internal focus group second in the cross over.
  Interventions: Other: Focus of Attention

INTERVENTIONS:
Other: Focus of Attention — Focus of attention instruction and feedback. Focus of attention refers to what people are thinking about during motor tasks. An external focus refers to thinking about an outside outcome or target. An internal focus of attention refers to thinking about how someone is moving their body.

SUMMARY:
The purpose of this study is to explore whether an external focus or internal focus of attention leads to improved motor performance and learning with increased use of the affected side during sit to stand in individuals post stroke. Focus of attention refers to what a person is thinking about during a task, with an internal focus being thinking about what one's body is doing and an external focus being thinking about a target or outcome in the environment. A second purpose is to determine whether improved symmetry in sit to stand carries over to gait symmetry in individuals post stroke.

DETAILED DESCRIPTION:
Participant demographics including age, gender, weight, and height will be collected. Self-selected gait speed, temporospatial gait parameters, and 5 Times Sit to Stand, will be collected at baseline, immediately after, during short term retention (20 minutes after training), and long term retention (one hour after training is completed). Gait speed and temporospatial parameters will be averaged across four passes over the GaitRite mat with participants being instructed to 'walk past the end of the mat at a normal comfortable pace'. The 5 Times Sit to Stand test will be completed from an 20" height and participants will be instructed, "Stand up and sit down 5 times as quickly as possible without using arms".

Participants will then be seated on a pressure mat placed on hi-lo table at a height where the participant's thigh is parallel to the floor, with an IMU marker on the manubrium. The participant's feet will be placed on an HR pressure mat at a comfortable width with toes being in line with one another. Tape marks will be placed at initial foot and buttocks position to allow for a consistent positioning throughout all trials. For baseline measurement, participants will perform sit to stand three times. During baseline, participants will be instructed to "please stand up without arms if possible". Immediately post training, during short term, and long term retention participants will be told, "using the strategy used during training, please stand up without using arms three times" and "please stand up normally". Average force under the affected side/average overall force during the sit to stand transition will be captured on the HR pressure mat located beneath the participants feet.

Participants will be categorized into groups based on stroke chronicity with those who have had a stroke within 6 months being placed in the subacute group and those with a stroke greater than 6 months being categorized in the chronic group. Within their stroke category they will be randomized into either the internal or external focus group using a random number generator. Each participant will perform 3 trials of sit to stand at baseline, short term, and long-term retention. During training, participants will perform sets of sit to stands with the mat at progressively lower heights, with differing cues based on group allocation. One set of sit to stands to 10 or form fatigue or RPE rating >16/20 will occur 30% above baseline, 20%, and 10% of the starting mat height. If participants are unable to complete 10 the number completed will be recorded for each trial. Two minute rest breaks will occur between each set or until the paricipant reports a rate of perceived exertion (RPE) of <11/20 on the Borg RPE scale.

Prior to training the participants will be given a demonstration. The external focus group will be told, "Stand up and sit down trying to keep the orange targets and the blue targets as close together as possible, like this." The internal focus group will be told, "Stand up and sit down trying to keep the R/L shoulder and R/L hip as far to the R/L as possible, like this." Participants will be asked to perform one repetition, "show me". Corrections will be given based on participant performance and group allocation.

During acquisition trials the external focus group will have foam circles taped to their lateral shoulder and lateral hip. Matching circles will be placed half the body width plus 10cm to their side in line with the feet. See figure 2. This distance will be determined by taking the girth in sitting. Participants will be instructed to 'bring the targets together as participants stand up. The internal focus group will be instructed to bring the left/right shoulder and hip as far to the left/right as possible. Feedback will be provided according to group allocation.

Center of pressure beneath the feet at the maximum lateral excursion towards the affected side, as well as the average throughout sit to stand will be analyzed at baseline, during acquisition trials, immediately after training, 20 minutes later, and 1 hour after training. Trunk alignment will also be captured at these same times with the IMU.

During the 20 minutes between the training and short term data collection participants will complete a post manipulation questionnaire regarding what participants were thinking about during sit to stand training. During the hour between short term and long-term retention participants will complete a general health questionnaire and the Montreal Cognitive Assessment (MOCA) to explore cognitive status.

One week later participants will return and complete the same protocol in the opposite group initially assigned. Both sessions should last less than two hours.

ELIGIBILITY:
Inclusion Criteria:

* Stroke >1 month
* Must be able to perform sit to stand from a standard height 20" chair without physical assistance
* Must be able to walk 20 feet with or without an assistive device at a contact guard to independent level
* Follow 3 step motor commands.

Exclusion Criteria:

* Contraversive pushing
* Neglect as evidenced by <44/54 on the star cancellation test
* Any orthopedic conditions that impact their ability to transition from sit to stand will be excluded from the study.
* Any other neurologic conditions that impact their ability to transition from sit to stand will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-10-07 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Center of pressure under their feet | Baseline
  HR Pressure mat - Symmetry under the feet will be measured using a 61.26 X 58.72 cm pedobarograph with a 48.8 X 44.7 cm active sensing area during the sit to stand transition. The mat has 3.9 sensors/cm2 with a 185 Hz scanning rate. The mat will be calibrated prior to the start of the study.
Center of pressure under their feet | Acquisition (one 1 hour training)
  HR Pressure mat - Symmetry under the feet will be measured using a 61.26 X 58.72 cm pedobarograph with a 48.8 X 44.7 cm active sensing area during the sit to stand transition. The mat has 3.9 sensors/cm2 with a 185 Hz scanning rate. The mat will be calibrated prior to the start of the study.
Center of pressure under their feet | Immediate Post (2 minutes after acquisition training)
  HR Pressure mat - Symmetry under the feet will be measured using a 61.26 X 58.72 cm pedobarograph with a 48.8 X 44.7 cm active sensing area during the sit to stand transition. The mat has 3.9 sensors/cm2 with a 185 Hz scanning rate. The mat will be calibrated prior to the start of the study.
Center of pressure under their feet | Short term (20 minutes after post data collection)
  HR Pressure mat - Symmetry under the feet will be measured using a 61.26 X 58.72 cm pedobarograph with a 48.8 X 44.7 cm active sensing area during the sit to stand transition. The mat has 3.9 sensors/cm2 with a 185 Hz scanning rate. The mat will be calibrated prior to the start of the study.
Center of pressure under their feet | Long term (one hour after post data collection)
  HR Pressure mat - Symmetry under the feet will be measured using a 61.26 X 58.72 cm pedobarograph with a 48.8 X 44.7 cm active sensing area during the sit to stand transition. The mat has 3.9 sensors/cm2 with a 185 Hz scanning rate. The mat will be calibrated prior to the start of the study.
Trunk alignment | Baseline
  IMU sensors -One Delsys inertial measurement units (IMUs) will be placed on the T1 spinous process to capture vertical trunk alignment throughout sit to stand.
Trunk alignment | Acquisition (one 1 hour training)
  IMU sensors -One Delsys inertial measurement units (IMUs) will be placed on the T1 spinous process to capture vertical trunk alignment throughout sit to stand.
Trunk alignment | Immediate Post (2 minutes after acquisition training)
  IMU sensors -One Delsys inertial measurement units (IMUs) will be placed on the T1 spinous process to capture vertical trunk alignment throughout sit to stand.
Trunk alignment | Short term (20 minutes after post data collection)
  IMU sensors -One Delsys inertial measurement units (IMUs) will be placed on the T1 spinous process to capture vertical trunk alignment throughout sit to stand.
Trunk alignment | Long term (one hour after post data collection)
  IMU sensors -One Delsys inertial measurement units (IMUs) will be placed on the T1 spinous process to capture vertical trunk alignment throughout sit to stand.
5 times sit to stand | Baseline
  Five Times Sit to Stand will also be an outcome measure used at baseline, immediately after training, during short term retention (20 min after training) and long term retention (1 hour after training).
5 times sit to stand | Immediate Post (2 minutes after acquisition training)
  Five Times Sit to Stand will also be an outcome measure used at baseline, immediately after training, during short term retention (20 min after training) and long term retention (1 hour after training).
5 times sit to stand | Short term (20 minutes after post data collection)
  Five Times Sit to Stand will also be an outcome measure used at baseline, immediately after training, during short term retention (20 min after training) and long term retention (1 hour after training).
5 times sit to stand | Long term (one hour after post data collection)
  Five Times Sit to Stand will also be an outcome measure used at baseline, immediately after training, during short term retention (20 min after training) and long term retention (1 hour after training).

SECONDARY OUTCOMES:
Gait symmetry | Baseline
  GaitRite - A 20'X 4' GAITRite will be used to gather gait speed and analyze spatial temporal aspects of gait. The GAITRite mat is an electronic walkway which uses pressure activated sensors to map out foot placement during gait using a quadrilateral blocking system. The walkway is made up of sensor pads, each of which has 2,304 sensors arranged in 48X48 grids. The measurements are provided using x,y coordinates and algorithms in the computer system use this information to group sensors into footprints. The mat has a spatial resolution of 1.27 cm and a spatial resolution accuracy of 1.27 cm. The mat will be set at 120 Hz sampling rate. All other parameters are fixed. GAITRite software will be used to collect percent of time spent in affected lower extremity stance compared to total stance time.
Gait symmetry | Immediate Post (2 minutes after acquisition training)
  GaitRite - A 20'X 4' GAITRite will be used to gather gait speed and analyze spatial temporal aspects of gait. The GAITRite mat is an electronic walkway which uses pressure activated sensors to map out foot placement during gait using a quadrilateral blocking system. The walkway is made up of sensor pads, each of which has 2,304 sensors arranged in 48X48 grids. The measurements are provided using x,y coordinates and algorithms in the computer system use this information to group sensors into footprints. The mat has a spatial resolution of 1.27 cm and a spatial resolution accuracy of 1.27 cm. The mat will be set at 120 Hz sampling rate. All other parameters are fixed. GAITRite software will be used to collect percent of time spent in affected lower extremity stance compared to total stance time.
Gait symmetry | Short term (20 minutes after post data collection)
  GaitRite - A 20'X 4' GAITRite will be used to gather gait speed and analyze spatial temporal aspects of gait. The GAITRite mat is an electronic walkway which uses pressure activated sensors to map out foot placement during gait using a quadrilateral blocking system. The walkway is made up of sensor pads, each of which has 2,304 sensors arranged in 48X48 grids. The measurements are provided using x,y coordinates and algorithms in the computer system use this information to group sensors into footprints. The mat has a spatial resolution of 1.27 cm and a spatial resolution accuracy of 1.27 cm. The mat will be set at 120 Hz sampling rate. All other parameters are fixed. GAITRite software will be used to collect percent of time spent in affected lower extremity stance compared to total stance time.
Gait symmetry | Long term (one hour after post data collection)
  GaitRite - A 20'X 4' GAITRite will be used to gather gait speed and analyze spatial temporal aspects of gait. The GAITRite mat is an electronic walkway which uses pressure activated sensors to map out foot placement during gait using a quadrilateral blocking system. The walkway is made up of sensor pads, each of which has 2,304 sensors arranged in 48X48 grids. The measurements are provided using x,y coordinates and algorithms in the computer system use this information to group sensors into footprints. The mat has a spatial resolution of 1.27 cm and a spatial resolution accuracy of 1.27 cm. The mat will be set at 120 Hz sampling rate. All other parameters are fixed. GAITRite software will be used to collect percent of time spent in affected lower extremity stance compared to total stance time.

CONTACTS AND LOCATIONS:
Locations (1):
- Western Carolina University, Cullowhee, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No